CLINICAL TRIAL: NCT02545244
Title: "Effectiveness of Black Tea Mouthwash on Plaque Formation:A Randomized Controlled Clinical Trial"
Brief Title: Effectiveness of Black Tea Mouthwash on Plaque Formation
Acronym: Blacktea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sri Hasanamba Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr. Smitha K.B, MDS Student in Periodontics, Sri Hasanamba Dental College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHDCH/2015-16/1107
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Gingivitis
Keywords: Gingivitis, Black Tea, Green Tea,Chlorhexidine, Biofilm,
MeSH Terms: conditions — Gingivitis | interventions — Tea

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Black Tea (Experimental): 0.5% Black Tea as Mouthwash, 5mL to be used twice daily for 30 seconds undiluted.
  Interventions: Dietary Supplement: Black Tea
- Green Tea (Active Comparator): 0.5% Green Tea as Mouthwash, 5mL to be used twice daily for 30 seconds undiluted.
  Interventions: Dietary Supplement: Green Tea
- Chlorhexidine (Active Comparator): 0.12% Chlorhexidine Mouthwash 5mL to be used twice daily.
  Interventions: Drug: 0.12% Chlorhexidine Mouthwash.

INTERVENTIONS:
Dietary Supplement: Black Tea — 0.5% Black Tea 5mL used as Mouthwash twice daily for two weeks after scaling of teeth.
  Arms: Black Tea
Dietary Supplement: Green Tea — 0.5% Green Tea 5mL used as Mouthwash twice daily for two weeks after scaling of teeth.
  Arms: Green Tea
Drug: 0.12% Chlorhexidine Mouthwash. — 5mL of 0.12% Chlorhexidine used as mouthwash twice daily for two weeks after scaling of teeth.
  Arms: Chlorhexidine

SUMMARY:
The study was conducted to measure the effectiveness of Black Tea in reducing the deposits on teeth. It also compares the effect between use of black tea mouthwash and green tea mouthwash to that of chlorhexidine in reducing plaque deposition on teeth in a two weeks long clinical trial among adults of 18-40 years of age.

DETAILED DESCRIPTION:
The study titled "Effectiveness of Black Tea Mouthwash on Plaque formation: A Randomized Controlled Clinical Trial" conducted at Department of Periodontics,during February 2015 till July 2015 included three interventional arms with 15 subjects each who had chronic generalized plaque-induced gingivitis. All subjects underwent scaling and randomly allocated into three groups as Black tea,Green tea and Chlorhexidine. Those in black tea, green tea and Chlorhexidine groups advised to rinse with 0.5% Black tea, 0.5% green tea and 0.12% Chlorhexidine aqueous based solutions for 30 seconds twice daily half an hour after brushing teeth respectively. Gingival Index (Loe and Silness 1963) and Plaque Index (Silness and Loe, 1964) recorded at baseline and 2 weeks after intervention in all subjects. Results were analyzed using SPSS Statistical software version 20.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old. subjects with at least 20 natural teeth. diagnosed with chronic generalized plaque induced gingivitis.

Exclusion Criteria:

* subjects with systemic illness. subjects on antibiotic in the previous six months. subjects with allergy to tea. subjects on medications with effect on periodontium (Eg:anti-osteoporotic drugs).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Plaque Index (Silness and Loe 1964) | two weeks
  Plaque Index at baseline and two weeks after scaling and use of mouthwash

SECONDARY OUTCOMES:
Gingival Index(Loe and Silness 1963) | two weeks
  Measure Gingival Index at baseline and two weeks after scaling and use of mouthwash

CONTACTS AND LOCATIONS:
Overall Officials: ShivaMurthy Ravindra, MDS, Principal Investigator — Sri Hasanamba Dental College and Hospital
Locations (1):
- Sri Hasanamba Dental College and Hospital, Hassan, Karnataka, India